CLINICAL TRIAL: NCT03266588
Title: A Multicenter, Open Label Long-Term Safety Study of BHV-3000 in the Acute Treatment of Migraine
Brief Title: Open Label Safety Study in Acute Treatment of Migraine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV3000-201
Record Dates: First submitted 2017-08-23; First posted 2017-08-30 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Migraine, With or Without Aura
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rimegepant (Experimental)
  Interventions: Drug: Rimegepant

INTERVENTIONS:
Drug: Rimegepant — 75 mg oral tablet
  Other Names: BHV-3000

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of BHV-3000 (rimegepant).

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with 2-8 moderate to severe migraines/month
* Age of onset of migraines prior to 50 years of age
* Migraine attacks, on average, lasting 4-72 hours if untreated
* Ability to distinguish migraine attacks from tension/cluster headaches
* Patients with contraindications for use of triptans may be included provided they meet all other study entry criteria

Key Exclusion Criteria:

* History of basilar migraine or hemiplegic migraine
* History of HIV disease
* History with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia.
* Uncontrolled hypertension or uncontrolled diabetes (however, patients can be included who have stable hypertension and /or diabetes for 3 months prior to screening
* History of gastric or small intestinal surgery or has a disease that causes malabsorption
* BMI ≥ 30
* HbA1c ≥ 6.5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3019 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (97):
- United States (97):
  - Central Research Associates, Inc, Birmingham, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Thunderbird Internal Medicine / Radiant Research, Inc, Glendale, Arizona
  - Neurological Physicians of Arizona, Tempe, Arizona
  - Clinical Research Consortium Arizona, Tempe, Arizona
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - Pharmacology Research Institute, Encino, California
  - eStudySite, La Mesa, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pacific Research Partners LLC, Oakland, California
  - National Research Institute, Panorama City, California
  - Optimus Medical Group, San Francisco, California
  - California Medical Clinic for Headache, Santa Monica, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Diablo Clinical Research, Inc, Walnut Creek, California
  - Clinical Trials of the Rockies, Denver, Colorado
  - AGA Clinical Trials, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Multi-Specialty Research Associates, Inc, Lake City, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - Ormond Medical Arts Pharmaceutical Research, Ormond Beach, Florida
  - Meridien Research, Tampa, Florida
  - Radiant Research, Inc., Atlanta, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Savannah Neurology Specialists, Savannah, Georgia
  - Christie Clinic, LLC, Champaign, Illinois
  - PMG Research of McFrland Clinic, Ames, Iowa
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Benchmark Research, Metairie, Louisiana
  - MedPharmics, LLC, Metairie, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Boston Clinical Trials, Inc., Boston, Massachusetts
  - NECCR Primacare Research, LLC, Fall River, Massachusetts
  - Milford Emergency Associates, Inc., Marlborough, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Clinical Research Insitute, Plymouth, Minnesota
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Meridian Clinical Research -Norfolk, Norfolk, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Clinical Research Consortium- Las Vegas, Las Vegas, Nevada
  - Hassman Research Institute, LLC, Berlin, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - United Medical Associates, Binghamton, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Radiant Research, Inc., Jamaica, New York
  - Central New York Clinical Research, Manlius, New York
  - Fieve Clinical Research, New York, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Montefiore Heachache Center, The Bronx, New York
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - PharmQuest, LLC, Greensboro, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Radiant Research, Inc., Cincinnati, Ohio
  - Radiant Research, Inc., Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Aventiv Research, Inc., Dublin, Ohio
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc, Salem, Oregon
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Fieve Clinical Research, Scranton, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Radiant Research, Inc., Anderson, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - FutureSearch Trials of Neurology, LP, Austin, Texas
  - Tekton Research- Austin, Austin, Texas
  - FutureSearch Trials of Neurology, LP, Dallas, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Texas Center for Drug Development, Houston, Texas
  - Red Star Research, LLC, Lake Jackson, Texas
  - FMC Science, Lampasas, Texas
  - PCP for Life, Magnolia, Texas
  - Research Across America - Mesquite, Mesquite, Texas
  - Doctors of Internal Medicine, LTD / Radiant Research Inc., Plano, Texas
  - DM Clinical Research, Tomball, Texas
  - J.Lewis Research Inc / Foothill Family Clinic South, Salt Lake City, Utah
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Women's:Health, Research & Gynecology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ailani J, Pavlovic J, Pixton GC, Fullerton T. Rimegepant safety and patient-reported outcomes among triptan-naive, triptan-using, and triptan-failure participants: Subgroup analysis of an open-label, multicenter study. Cephalalgia. 2025 Jul;45(7):3331024251343309. doi: 10.1177/03331024251343309. Epub 2025 Jul 9. PMID 40629887
- [Derived] Kudrow D, Hutchinson S, Pixton GC, Fullerton T. Safety of Rimegepant in Adults with Migraine and Anxiety, Depression, or Using Antidepressants: Analysis of a Multicenter, Long-Term, Open-Label Study. Pain Ther. 2025 Feb;14(1):237-255. doi: 10.1007/s40122-024-00675-6. Epub 2024 Nov 9. PMID 39520634
- [Derived] True D, Mullin K, Croop R. Safety of Rimegepant in Adults with Migraine and Cardiovascular Risk Factors: Analysis of a Multicenter, Long-Term, Open-Label Study. Pain Ther. 2024 Oct;13(5):1203-1218. doi: 10.1007/s40122-024-00626-1. Epub 2024 Jul 10. PMID 38985436
- [Derived] Fullerton T, Pixton G. Long-Term Use of Rimegepant 75 mg for the Acute Treatment of Migraine is Associated with a Reduction in the Utilization of Select Analgesics and Antiemetics. J Pain Res. 2024 May 15;17:1751-1760. doi: 10.2147/JPR.S456006. eCollection 2024. PMID 38764606
- [Derived] Croop R, Berman G, Kudrow D, Mullin K, Thiry A, Lovegren M, L'Italien G, Lipton RB. A multicenter, open-label long-term safety study of rimegepant for the acute treatment of migraine. Cephalalgia. 2024 Apr;44(4):3331024241232944. doi: 10.1177/03331024241232944. PMID 38659334
- [Derived] Johnston K, Harris L, Powell L, Popoff E, Coric V, L'Italien G, Schreiber CP. Monthly migraine days, tablet utilization, and quality of life associated with Rimegepant - post hoc results from an open label safety study (BHV3000-201). J Headache Pain. 2022 Jan 17;23(1):10. doi: 10.1186/s10194-021-01378-5. PMID 35038983
- [Derived] Johnston KM, L'Italien G, Popoff E, Powell L, Croop R, Thiry A, Harris L, Coric V, Lipton RB. Mapping Migraine-Specific Quality of Life to Health State Utilities in Patients Receiving Rimegepant. Adv Ther. 2021 Oct;38(10):5209-5220. doi: 10.1007/s12325-021-01897-2. Epub 2021 Aug 29. PMID 34455556
- [Derived] Mullin K, Kudrow D, Croop R, Lovegren M, Conway CM, Coric V, Lipton RB. Potential for treatment benefit of small molecule CGRP receptor antagonist plus monoclonal antibody in migraine therapy. Neurology. 2020 May 19;94(20):e2121-e2125. doi: 10.1212/WNL.0000000000008944. Epub 2020 Jan 13. PMID 31932515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 103 centers in the United States.
Pre-assignment Details: A total of 3019 participants were screened for this open-label study. A total of 2867 participants entered the observational period, and 1908 participants subsequently enrolled in the long-term treatment period of whom 1800 received treatment. A total of 807 participants failed screening mainly due to failure to meet eligibility criteria.
Groups:
- PRN (2-8) Group: To meet entry criteria, these participants had to have a self-reported historical rate of 2 to 8 moderate to severe migraine attacks per month preceding enrollment in the group. Participants were allowed to dose as needed (PRN), up to 1 tablet per calendar day, with 75 mg of rimegepant tablet. While on-treatment, participants were allowed to treat migraine attacks of any severity (mild, moderate, or severe) for a planned duration up to 52 weeks.
- PRN (9-14) Group: To meet entry criteria, these participants had to have a self-reported historical rate of 9 to 14 moderate to severe migraine attacks per month preceding enrollment in the group. Participants were allowed to dose as needed (PRN), up to 1 tablet per calendar day, with 75 mg of rimegepant tablet. While on-treatment, participants were allowed to treat migraine attacks of any severity (mild, moderate, or severe) for a planned duration up to 52 weeks.
- Scheduled EOD + PRN Group: To meet entry criteria, these participants had to have a self-reported historical rate of 4 to 14 moderate to severe migraine attacks per month preceding enrollment in the group. Participants were allowed to dose every other day (EOD); on the days that participants were not scheduled for dosing, the participants were allowed to dose on an as-needed basis (PRN), up to 1 tablet per calendar day, with 75 mg of rimegepant tablet. While on-treatment, participants were allowed to treat migraine attacks of any severity (mild, moderate, or severe) for a planned duration up to 12 weeks.
Period: Observational Period
Arm/Group | PRN (2-8) Group | PRN (9-14) Group | Scheduled EOD + PRN Group
Started (Number includes participants who entered the Observation Period.) | 1605 | 786 | 476
Completed | 1089 | 511 | 308
Not Completed | 516 | 275 | 168
Not completed — Screen Failure: Eligibility Criteria | 439 | 228 | 140
Not completed — Withdrawal by Subject | 44 | 22 | 13
Not completed — Non-compliance | 18 | 12 | 10
Not completed — Lost to Follow-up | 8 | 12 | 4
Not completed — Eligibility Failure- Baseline Lab Values | 3 | 1 | 0
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Other Reasons | 3 | 0 | 1
Period: Long-term Treatment Period
Arm/Group | PRN (2-8) Group | PRN (9-14) Group | Scheduled EOD + PRN Group
Started | 1089 | 511 | 308
Treated | 1033 | 481 | 286
Completed | 683 | 271 | 243
Not Completed | 406 | 240 | 65
Not completed — Adverse Event | 33 | 17 | 8
Not completed — Lack of Efficacy | 41 | 31 | 5
Not completed — Lost to Follow-up | 39 | 37 | 8
Not completed — Non-Compliance | 126 | 57 | 7
Not completed — Pregnancy | 11 | 5 | 0
Not completed — Protocol Deviation | 17 | 10 | 4
Not completed — Screen Failure: Eligibility Criteria | 33 | 17 | 17
Not completed — Withdrawal by Subject | 100 | 63 | 16
Not completed — No Migraine Treated by Week 8 Visit | 1 | 2 | 0
Not completed — Other Reasons | 5 | 0 | 0
Not completed — Positive Sheehan-STS Score > 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was performed on treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | PRN (2-8) Group | PRN (9-14) Group | Scheduled EOD + PRN Group | Total
Number analyzed (Participants) | 1033 | 481 | 286 | 1800
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (11.79) | 42.4 (12.41) | 41.1 (12.69) | 43.1 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 917 | 444 | 248 | 1609
  Male | 116 | 37 | 38 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99 | 54 | 24 | 177
  Not Hispanic or Latino | 934 | 427 | 262 | 1623
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 2 | 10
  Asian | 16 | 7 | 9 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 2 | 5
  Black or African American | 149 | 66 | 35 | 250
  White | 847 | 394 | 234 | 1475
  More than one race | 17 | 7 | 4 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1033 | 481 | 286 | 1800

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With SAEs and AEs Leading to Discontinuation During the Treatment Period
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition on-treatment in a patient or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. An SAE was defined as any event that met any of the following criteria: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received rimegepant; other important medical events that may not have resulted in death, be life-threatening, or required hospitalization, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention.
Time Frame: PRN (2-8) and PRN (9-14) groups: Up to 52 weeks; Scheduled EOD + PRN group: Up to 12 weeks
Population: The analysis was performed on treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | PRN (2-8) Group | PRN (9-14) Group | Scheduled EOD + PRN Group
Number analyzed (Participants) | 1033 | 481 | 286
Participants
  Overall number of participants with at least 1 AE | 664 | 315 | 109
  AE ≥5%-Upper respiratory tract infection | 108 | 38 | 12
  Mild-Upper respiratory tract infection | 56 | 21 | 8
  Moderate-Upper respiratory tract infection | 51 | 17 | 4
  Severe-Upper respiratory tract infection | 1 | 0 | 0
  AE ≥5%-Nasopharyngitis | 72 | 41 | 9
  Mild-Nasopharyngitis | 53 | 28 | 7
  Moderate-Nasopharyngitis | 19 | 13 | 2
  AE ≥5%-Sinusitis | 57 | 28 | 7
  Mild-Sinusitis | 26 | 19 | 5
  Moderate-Sinusitis | 30 | 9 | 2
  Severe-Sinusitis | 1 | 0 | 0
  SAEs | 28 | 16 | 3
  AEs leading to discontinuation | 24 | 16 | 8

2. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities During the Treatment Period
Description: Clinically significant laboratory abnormalities were defined as Grade 3 to 4 on-treatment laboratory test results according to numeric laboratory test criteria found in Common Technical Criteria for Adverse Events (CTCAE) Version 5.0 (2017) if available; otherwise, according to Division of Acquired Immune Deficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1 (2017) for Glucose, LDL-Cholesterol, Uric Acid, and Urinalysis. Laboratory test groups of clinical interest included hematology, serum chemistry, and urinalysis. Participants must have had a non-missing measurement in the on-treatment period to be included for a given parameter.
Time Frame: PRN (2-8) and PRN (9-14) groups: Up to 52 weeks: Scheduled EOD + PRN group: Up to 12 weeks
Population: The analysis was performed on treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | PRN (2-8) Group | PRN (9-14) Group | Scheduled EOD + PRN Group
Number analyzed (Participants) | 1033 | 481 | 286
Participants
  Alanine Aminotransferase (ALT): number analyzed (Participants) | 1017 | 466 | 279
  Alanine Aminotransferase (ALT) | 3 | 2 | 0
  Aspartate Aminotransferase (AST): number analyzed (Participants) | 1017 | 466 | 279
  Aspartate Aminotransferase (AST) | 4 | 2 | 0
  Albumin: number analyzed (Participants) | 996 | 458 | 276
  Albumin | 0 | 0 | 0
  Alkaline Phosphatase: number analyzed (Participants) | 1017 | 466 | 279
  Alkaline Phosphatase | 0 | 0 | 0
  Bicarbonate: number analyzed (Participants) | 996 | 458 | 276
  Bicarbonate | 0 | 0 | 0
  Bilirubin: number analyzed (Participants) | 1017 | 466 | 279
  Bilirubin | 0 | 0 | 0
  Calcium, Low: number analyzed (Participants) | 996 | 458 | 276
  Calcium, Low | 0 | 0 | 0
  Calcium, High: number analyzed (Participants) | 996 | 458 | 276
  Calcium, High | 0 | 0 | 0
  Cholesterol: number analyzed (Participants) | 899 | 387 | 260
  Cholesterol | 0 | 0 | 0
  Creatine Kinase: number analyzed (Participants) | 996 | 458 | 276
  Creatine Kinase | 16 | 10 | 3
  Creatinine: number analyzed (Participants) | 996 | 458 | 276
  Creatinine | 1 | 0 | 0
  Glomerular Filtration Rate, Estimated: number analyzed (Participants) | 996 | 458 | 276
  Glomerular Filtration Rate, Estimated | 1 | 0 | 0
  Glucose, Low: number analyzed (Participants) | 996 | 458 | 276
  Glucose, Low | 1 | 1 | 1
  Glucose, High: number analyzed (Participants) | 996 | 458 | 276
  Glucose, High | 10 | 1 | 0
  LDL-cholesterol: number analyzed (Participants) | 899 | 387 | 260
  LDL-cholesterol | 31 | 15 | 2
  Lactate Dehydrogenase: number analyzed (Participants) | 996 | 458 | 276
  Lactate Dehydrogenase | 0 | 0 | 0
  Potassium, Low: number analyzed (Participants) | 996 | 458 | 276
  Potassium, Low | 2 | 0 | 0
  Potassium, High: number analyzed (Participants) | 996 | 458 | 276
  Potassium, High | 3 | 2 | 0
  Sodium, Low: number analyzed (Participants) | 996 | 458 | 276
  Sodium, Low | 1 | 0 | 0
  Sodium, High: number analyzed (Participants) | 996 | 458 | 276
  Sodium, High | 0 | 0 | 0
  Triglycerides: number analyzed (Participants) | 899 | 387 | 260
  Triglycerides | 1 | 1 | 3
  Uric Acid: number analyzed (Participants) | 996 | 458 | 276
  Uric Acid | 0 | 0 | 0
  Hemoglobin: number analyzed (Participants) | 995 | 458 | 276
  Hemoglobin | 2 | 1 | 0
  Lymphocytes, Low: number analyzed (Participants) | 995 | 458 | 276
  Lymphocytes, Low | 0 | 0 | 0
  Lymphocytes, High: number analyzed (Participants) | 995 | 458 | 276
  Lymphocytes, High | 0 | 1 | 0
  Neutrophils: number analyzed (Participants) | 995 | 458 | 276
  Neutrophils | 4 | 0 | 1
  Platelets: number analyzed (Participants) | 995 | 457 | 276
  Platelets | 0 | 0 | 0
  White Blood Cells: number analyzed (Participants) | 995 | 458 | 276
  White Blood Cells | 0 | 0 | 0
  Urine Erythrocytes: number analyzed (Participants) | 263 | 113 | 76
  Urine Erythrocytes | 0 | 0 | 0
  Urine Glucose: number analyzed (Participants) | 664 | 308 | 256
  Urine Glucose | 10 | 2 | 0
  Urine Protein: number analyzed (Participants) | 664 | 308 | 256
  Urine Protein | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Elevations of AST or ALT > 3 x Upper Limit of Normal (ULN) Concurrent With Total Bilirubin > 2 x ULN During the Treatment Period
Description: Elevations of on-treatment AST or ALT > 3 x ULN concurrent with total bilirubin > 2 x ULN were defined as elevations on the same collection date.
Time Frame: PRN (2-8) and PRN (9-14) groups: Up to 52 weeks; Scheduled EOD + PRN group: Up to 12 weeks
Population: The analysis was performed on treated participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PRN (2-8) Group | PRN (9-14) Group | Scheduled EOD + PRN Group
Number analyzed (Participants) | 1033 | 481 | 286
Percentage of participants | 0.1 [0.00 to 0.60] | 0 [0.00 to 0.96] | 0 [0.00 to 1.60]

4. Secondary Outcome: Number of Participants With Hepatic-related AEs and Hepatic-related AEs Leading to Discontinuation During the Treatment Period
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition on-treatment in a patient or clinical investigation patient administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. Hepatic AEs were defined as all on-treatment PTs under the "Hepatic Disorders" Standardized Medical Dictionary (Version 21.1) for Regulatory Activities Query (SMQ), except those PTs in the "Congenital, Familial, Neonatal and Genetic Disorders of the Liver" SMQ.
Time Frame: PRN (2-8) and PRN (9-14) groups: Up to 52 weeks; Scheduled EOD + PRN group: Up to 12 weeks
Population: The analysis was performed on treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | PRN (2-8) Group | PRN (9-14) Group | Scheduled EOD + PRN Group
Number analyzed (Participants) | 1033 | 481 | 286
Participants
  Hepatic-related AE | 16 | 10 | 0
  Hepatic-related AE leading to discontinuation | 3 | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from start of study drug treatment up to 52 weeks
Description: The analysis was performed on treated participants.
Groups:
- Scheduled EOD + PRN Group: To meet entry criteria, these participants had to have a self-reported historical rate of 4 to 14 moderate to severe migraine attacks per month preceding enrollment in the group. Participants were allowed to dose every other day (EOD); on the days that participants were not scheduled for dosing, the participants were allowed to dose on an as-needed basis (PRN), up to 1 tablet per calendar day, with 75 mg of rimegepant tablet. While ontreatment, participants were allowed to treat migraine attacks of any severity (mild, moderate, or severe) for a planned duration up to 12 weeks.
Arm/Group | PRN (2-8) Group | PRN (9-14) Group | Scheduled EOD + PRN Group
All-Cause Mortality (participants affected / at risk) | 0/1033 | 0/481 | 0/286
Serious Adverse Events (participants affected / at risk) | 28/1033 | 16/481 | 3/286
Other Adverse Events (participants affected / at risk) | 224/1033 | 100/481 | 27/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRN (2-8) Group (N=1033) | PRN (9-14) Group (N=481) | Scheduled EOD + PRN Group (N=286)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 3 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Viral sepsis (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0
Hemiplegic migraine (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PRN (2-8) Group (N=1033) | PRN (9-14) Group (N=481) | Scheduled EOD + PRN Group (N=286)
Nasopharyngitis (Infections and infestations) | 72 | 41 | 9
Sinusitis (Infections and infestations) | 57 | 28 | 7
Upper respiratory tract infection (Infections and infestations) | 108 | 38 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03266588/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT03266588/SAP_001.pdf